CLINICAL TRIAL: NCT04209634
Title: An Open-Label Efficacy and Safety Study of Pozelimab in Patients With CD55-Deficient Protein-Losing Enteropathy (CHAPLE Disease)
Brief Title: Open-Label Efficacy and Safety Study of Pozelimab in Patients With CD55-Deficient Protein-Losing Enteropathy (CHAPLE Disease)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R3918-PLE-1878
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Results first posted 2023-10-30 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: CD55-deficient Protein-losing Enteropathy; CHAPLE
Keywords: CD55-deficient PLE; complement hyperactivation, angiopathic thrombosis, protein-losing enteropathy (CHAPLE disease)
MeSH Terms: conditions — Protein-Losing Enteropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active PLE (Experimental): Patients aged 1 year and older with a clinical diagnosis of CD55-deficient PLE disease
  Interventions: Drug: Pozelimab

INTERVENTIONS:
Drug: Pozelimab — Single loading intravenous (IV) dose on day 1, then fixed doses sub-cutaneous (SC) (based on body weight) QW (±2 days) over the treatment period.
  Other Names: REGN3918

SUMMARY:
The primary objective of the study is to determine the effect of pozelimab on active CD55-deficient protein-losing enteropathy (PLE; CHAPLE).

The secondary objectives of the study are:

* To evaluate the safety and tolerability of pozelimab in patients with CD55-deficient PLE disease
* To evaluate the effect of pozelimab on CD55-deficient PLE (both patients with active disease at baseline and those with inactive disease on eculizumab, switching to pozelimab)
* To determine the effects of pozelimab on albumin and other serum proteins (total protein, immunoglobulins)
* To determine the effects of pozelimab on ascites
* To determine the effects of pozelimab on stool consistency
* To determine the effect of pozelimab on health-related quality of life
* To determine the effect of pozelimab on lab abnormalities observed in CD55-deficient PLE such as hypertriglyceridemia, thrombocytosis, and hypovitaminosis B12
* To describe the effects of pozelimab on the sparing of concomitant medications and reduction in hospitalization days
* To determine the effects of pozelimab on growth
* To characterize the concentration of pozelimab in patients with CD55-deficient PLE
* To assess the incidence of treatment-emergent ADA for pozelimab in patients with CD55-deficient PLE disease

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical diagnosis of CD55-deficient PLE/CHAPLE disease (based on a history of PLE), confirmed by biallelic CD55 loss-of-function mutation detected by genotype analysis
* Active disease as defined by the protocol or inactive disease on eculizumab therapy (and whose treating physician has the expectation of future access to renewed eculizumab treatment should this be required), and is willing to discontinue eculizumab during screening and start pozelimab at baseline with no eculizumab wash-out

Key Exclusion Criteria:

* History of meningococcal infection
* No documented meningococcal vaccination within 3 years prior to screening and patient unwilling to undergo vaccination during the study
* No documented vaccination for Haemophilus influenzae and Streptococcus pneumoniae if applicable based on local practice or guidelines prior to screening and patient unwilling to undergo vaccination during the study if required per local practice or guidelines
* Presence of a concomitant disease that leads to hypoproteinemia at the time of starting pozelimab
* A concomitant disease that leads to secondary intestinal lymphangiectasia such as a fontan procedure for congenital heart disease

Note: Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2024-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (3):
- Regeneron Research Site, Bethesda, Maryland, United States
- Regeneron Research Site, Pathum Wan, Bangkok, Thailand
- Regeneron Research Site, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., FDA, EMA, PMDA, etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/

REFERENCES:
- [Derived] Litcher-Kelly L, Ozen A, Ollis S, Feldman HB, Yaworsky A, Medrano P, Chongsrisawat V, Perlee L, Walker M, Pradeep S, Turner-Bowker DM, Kurolap A, Adiv OE, Lenardo MJ, Harari OA, Jalbert JJ. The patient experience of CHAPLE disease: results from interviews conducted as part of a clinical trial for an ultra-rare condition. Orphanet J Rare Dis. 2025 Feb 11;20(1):68. doi: 10.1186/s13023-024-03436-y. PMID 39934837
- [Derived] Litcher-Kelly L, Ozen A, Ollis S, Feldman HB, Yaworsky A, Medrano P, Chongsrisawa V, Brackin T, Perlee L, Walker M, Pradeep S, Lenardo MJ, Harari OA, Jalbert JJ. Pozelimab for CHAPLE disease: results from in-trial interviews and clinical outcome assessments. Orphanet J Rare Dis. 2024 Aug 8;19(1):290. doi: 10.1186/s13023-024-03277-9. PMID 39118150
- [Derived] Ozen A, Chongsrisawat V, Sefer AP, Kolukisa B, Jalbert JJ, Meagher KA, Brackin T, Feldman HB, Baris S, Karakoc-Aydiner E, Ergelen R, Fuss IJ, Moorman H, Suratannon N, Suphapeetiporn K, Perlee L, Harari OA, Yancopoulos GD, Lenardo MJ; Pozelimab CHAPLE Working Group. Evaluating the efficacy and safety of pozelimab in patients with CD55 deficiency with hyperactivation of complement, angiopathic thrombosis, and protein-losing enteropathy disease: an open-label phase 2 and 3 study. Lancet. 2024 Feb 17;403(10427):645-656. doi: 10.1016/S0140-6736(23)02358-9. Epub 2024 Jan 23. PMID 38278170
- See also: A Plain Language Summary is available on TrialSummaries.com — https://www.trialsummaries.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 11 participants were screened for this study. Of these, 1 participant did not meet inclusion/exclusion criteria, and 10 were assigned to study treatment.
Groups:
- Pozelimab Injection: Participants received a single loading dose of pozelimab 30 milligrams per kilogram (mg/kg) intravenous (IV) injection on day 1, followed by weekly subcutaneous (SC) injection as maintenance dosing of 125 mg for body weight less than (<) 10 kilograms (kg), 200 mg for greater than or equal to (>=) 10 kg and <20 kg, 350 mg for >=20 kg and <40 kg, 500 mg for >=40 kg and <60 kg, and 800 mg for >=60 kg over the treatment period.
Period: Overall Study
Arm/Group | Pozelimab Injection
Started | 10
Completed (Completed study) | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all enrolled participants who received the study drug.
Groups:
- Pozelimab Injection: Participants received a single loading dose of pozelimab 30 mg/kg IV injection on day 1, followed by weekly SC injection as maintenance dosing of 125 mg for body weight <10 kg, 200 mg for >=10 kg and <20 kg, 350 mg for >=20 kg and <40 kg, 500 mg for >=40 kg and <60 kg, and 800 mg for >=60 kg over the treatment period.
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.3 (4.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Active Disease at Baseline Who Achieved Normalization of Serum Albumin and Improvement in Prespecified Clinical Outcomes at Week 24
Description: Normalization of serum albumin was defined as serum albumin within the normal range at least 70 percent (%) of measurements between weeks 12 and 24, and no single albumin measurement of <2.5 grams per deciliter (g/dL) between weeks 12 and 24, and no requirement for albumin infusion between weeks 12 and 24. Improvement in the following 4 prespecified clinical outcomes that were evaluable for improvement at baseline, without worsening of the others: Daily bowel movement frequency, the presence and severity of facial edema (physician-reported), the presence and severity of peripheral edema (physician-reported), and the participant/caregiver assessment of frequency of problematic abdominal pain. Percentage of participants with active disease at baseline who achieved normalization of serum albumin and improvement in prespecified clinical outcomes at Week 24 were reported.
Time Frame: At Week 24
Population: The FAS included all enrolled participants who received the study drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
percentage of participants | 100 [74.1 to 100]

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Severity of TEAEs
Description: TEAEs are defined as AEs that developed or worsened during the on-treatment period. The on-treatment period is defined as the time from first dose of investigational product up to 21 weeks after the last dose of investigational product. Severity of TEAEs was graded according to the following scale: Mild: Does not interfere in a significant manner with the patient's normal functioning level, Moderate: Produces some impairment of functioning but is not hazardous to health and Severe: Produces significant impairment of functioning or incapacitation and is a definite hazard to the participants health.
Time Frame: From start of study drug administration up to approximately 144 weeks
Population: The safety analysis set included all enrolled participants who received the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
Participants
  Participants with TEAEs | 10
  Participants with mild severity | 3
  Participants with moderate severity | 5
  Participants with severe severity | 2

3. Secondary Outcome: Number of Participants With Improvement in Most Bothersome Signs and Symptoms at Week 24
Description: Improvement in most bothersome sign/symptom determined using semi-structured concept elicitation interview, from 'core' clinical endpoints of frequency of bowel movements, peripheral edema, facial edema, abdominal pain frequency, nausea, vomiting, stool consistency.
Time Frame: At Week 24
Population: FAS included all enrolled participants who received the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
Participants | 10

4. Secondary Outcome: Number of Bowel Movements Per Day Based on a 1-week Average up to Week 24
Description: Daily bowel movements captured by e-diary. The number of bowel movements per day was calculated each week of the study. It was based on a 1-week average and calculated as the sum of the number of bowel movements in a given week divided by the number of days with non-missing bowel movement frequency data. If more than 3 days of bowel movement data was missing in a given week, bowel movement frequency data was considered missing for that week.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11,12,13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23 and 24
Population: FAS included all enrolled participants who received the study drug. Here, "number analyzed" signifies those participants who were evaluable for specified timepoints in categories.
Measure: Median (Full Range); unit: Bowel movements per day
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
Bowel movements per day
  Baseline | 1.64 [0.5 to 3.4]
  Week 1 | 1.13 [0.3 to 3.0]
  Week 2 | 1.36 [0.7 to 3.4]
  Week 3 | 1.43 [0.7 to 2.4]
  Week 4 | 1.50 [0.8 to 2.6]
  Week 5 | 1.57 [0.5 to 2.3]
  Week 6 | 1.21 [0.6 to 3.0]
  Week 7 | 1.21 [0.3 to 2.5]
  Week 8 | 1.07 [0.2 to 2.3]
  Week 9 | 1.00 [0.3 to 2.0]
  Week 10 | 1.00 [0.5 to 1.7]
  Week 11 | 1.00 [0.2 to 2.0]
  Week 12 | 0.79 [0.0 to 1.9]
  Week 13 | 0.93 [0.1 to 2.3]
  Week 14 | 0.93 [0.3 to 2.1]
  Week 15 | 1.07 [0.3 to 2.3]
  Week 16 | 1.10 [0.4 to 2.0]
  Week 17 | 1.13 [0.3 to 2.0]
  Week 18 | 1.00 [0.0 to 1.9]
  Week 19 | 1.00 [0.3 to 1.9]
  Week 20 | 0.83 [0.2 to 2.1]
  Week 21 | 1.00 [0.5 to 1.7]
  Week 22: number analyzed (Participants) | 9
  Week 22 | 0.83 [0.4 to 1.7]
  Week 23 | 0.86 [0.5 to 1.8]
  Week 24 | 0.90 [0.3 to 2.0]

5. Secondary Outcome: Number of Days Per Week With >=1 Bowel Movement of Loose/Watery Stool Consistency at Week 24
Description: The number of days per week with >=1 loose/watery bowel movement, is calculated each week of the study as the sum of the number of days with >=1 loose/watery bowel movement in a given week divided by the number of days with non-missing stool consistency data and then multiplied by 7, is presented. If more than 3 days of stool consistency data was missing in a given week, stool consistency data was considered missing for that week.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11,12,13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23 and 24
Population: FAS included all enrolled participants who received any study drug. Here, "number analyzed" signifies those participants who were evaluable for specified timepoints in categories.
Measure: Median (Full Range); unit: Days per week
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
Days per week
  Baseline | 2.00 [0.0 to 7.0]
  Week 1 | 0.50 [0.0 to 5.0]
  Week 2 | 0.00 [0.0 to 2.0]
  Week 3 | 0.00 [0.0 to 3.0]
  Week 4 | 0.00 [0.0 to 4.0]
  Week 5 | 0.00 [0.0 to 5.0]
  Week 6 | 1.20 [0.0 to 5.0]
  Week 7 | 0.50 [0.0 to 2.8]
  Week 8 | 0.50 [0.0 to 3.0]
  Week 9 | 0.50 [0.0 to 3.0]
  Week 10 | 0.00 [0.0 to 4.0]
  Week 11 | 1.00 [0.0 to 2.3]
  Week 12 | 0.00 [0.0 to 2.3]
  Week 13 | 0.00 [0.0 to 4.0]
  Week 14 | 1.58 [0.0 to 4.7]
  Week 15 | 1.00 [0.0 to 7.0]
  Week 16 | 0.00 [0.0 to 5.8]
  Week 17 | 1.28 [0.0 to 5.6]
  Week 18 | 0.50 [0.0 to 7.0]
  Week 19 | 0.00 [0.0 to 5.0]
  Week 20 | 0.00 [0.0 to 5.0]
  Week 21 | 0.00 [0.0 to 6.0]
  Week 22: number analyzed (Participants) | 9
  Week 22 | 0.00 [0.0 to 6.0]
  Week 23 | 0.00 [0.0 to 6.0]
  Week 24 | 0.00 [0.0 to 5.6]

6. Secondary Outcome: Number of Participants With Abdominal Ascites at Week 24
Description: The measurement of abdominal ascites (excess abdominal fluid) was based on abdominal circumference. Abdominal circumference was measured regardless of the physician's assessment of the presence or absence of ascites.
Time Frame: Baseline up to Week 24
Population: FAS included all enrolled participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
Participants | 1

7. Secondary Outcome: Absolute Value of Albumin at Specified Timepoints up to Week 24
Description: Blood samples were collected from participants at defined time points for the assessment of albumin. Absolute value of albumin at specified timepoints was reported.
Time Frame: Baseline, Day 2, Weeks 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22 and 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
g/dL
  Baseline | 2.160 (0.5296)
  Day 2: number analyzed (Participants) | 9
  Day 2 | 2.267 (0.4000)
  Week 1: number analyzed (Participants) | 9
  Week 1 | 3.311 (0.4485)
  Week 2: number analyzed (Participants) | 9
  Week 2 | 3.589 (0.4428)
  Week 3: number analyzed (Participants) | 8
  Week 3 | 4.025 (0.3955)
  Week 4: number analyzed (Participants) | 9
  Week 4 | 4.167 (0.3841)
  Week 6: number analyzed (Participants) | 9
  Week 6 | 4.411 (0.7026)
  Week 8: number analyzed (Participants) | 8
  Week 8 | 4.188 (0.3137)
  Week 10: number analyzed (Participants) | 9
  Week 10 | 4.322 (0.2279)
  Week 12: number analyzed (Participants) | 8
  Week 12 | 4.288 (0.2748)
  Week 14: number analyzed (Participants) | 8
  Week 14 | 4.363 (0.2615)
  Week 16: number analyzed (Participants) | 9
  Week 16 | 4.367 (0.3674)
  Week 18: number analyzed (Participants) | 9
  Week 18 | 4.344 (0.2555)
  Week 20 | 4.449 (0.2539)
  Week 22: number analyzed (Participants) | 9
  Week 22 | 4.422 (0.2906)
  Week 24: number analyzed (Participants) | 9
  Week 24 | 4.544 (0.2603)

8. Secondary Outcome: Absolute Values of Protein, and Immunoglobulin G (IgG) at Baseline and Week 24
Description: Blood samples were collected from participants at defined time points for the assessment of protein and IgG. Absolutes values of protein and IgG measured as g/L at baseline and Week 24 was reported.
Time Frame: Baseline, Week 24
Population: The safety analysis set included all enrolled participants who received the study drug. Here, "number analyzed" signifies those participants who were evaluable for specified timepoints in categories.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
g/L
  Protein at Baseline | 37.50 (6.996)
  Protein at Week 24: number analyzed (Participants) | 9
  Protein at Week 24 | 72.22 (4.969)
  IgG at Baseline | 2.183 (0.9103)
  IgG at Week 24: number analyzed (Participants) | 8
  IgG at Week 24 | 11.301 (2.0503)

9. Secondary Outcome: Absolute Values of Immunoglobulin (Ig), Immunoglobulin M (IgM), and Immunoglobulin A (IgA) at Baseline and Week 24
Description: Blood samples were collected from participants at defined time points for the assessment of Ig, IgM and IgA. Absolute value of Ig, IgM and IgA measured as mg/dL at baseline and Week 24 was reported.
Time Frame: Baseline, Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
mg/dL
  Ig at Baseline | 318.2 (113.36)
  Ig at Week 24: number analyzed (Participants) | 8
  Ig at Week 24 | 1430.1 (263.36)
  IgM at Baseline | 52.9 (28.36)
  IgM at Week 24: number analyzed (Participants) | 8
  IgM at Week 24 | 180.3 (74.81)
  IgA at Baseline | 47.0 (18.51)
  IgA at Week 24: number analyzed (Participants) | 8
  IgA at Week 24 | 119.8 (52.46)

10. Secondary Outcome: Absolute Values of Vitamin B12 at Baseline and Week 24
Description: Blood samples were collected from participants at defined time points for the assessment of vitamin B12. Absolute values of vitamin B12 at baseline and Week 24 was reported.
Time Frame: Baseline, Week 24
Population: The safety analysis set included all enrolled participants who received the study drug. Here, "overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: picomoles per liter (pmol/L)
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 8
picomoles per liter (pmol/L)
  Baseline | 158.5 (52.32)
  Week 24 | 383.1 (102.73)

11. Secondary Outcome: Absolute Values of Iron and Unsaturated Iron Binding Capacity at Baseline and Week 24
Description: Blood samples were collected from participants at defined time points for the assessment of iron indices. Absolute values of unsaturated iron and unsaturated iron binding capacity measured as micromoles per liter (mcmol/L) at baseline and Week 24 was reported.
Time Frame: Baseline, Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mcmol/L
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
mcmol/L
  Iron at Baseline | 3.40 (1.478)
  Iron at Week 24: number analyzed (Participants) | 8
  Iron at Week 24 | 7.38 (5.036)
  Unsaturated Binding Capacity at Baseline | 38.24 (12.357)
  Unsaturated Iron Binding Capacity at Week 24: number analyzed (Participants) | 8
  Unsaturated Iron Binding Capacity at Week 24 | 73.95 (12.049)

12. Secondary Outcome: Absolute Values of Vitamin B9 up to Week 24
Description: Absolute Values of Vitamin B9 - Central Lab
Time Frame: Baseline up to Week 24
Population: Number of participants based on the total in the safety analysis set (SAF)
Measure: Mean (Standard Deviation); unit: nanomoles per liter (nmol/L)
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
nanomoles per liter (nmol/L)
  Week 1 | 17.80 (15.017)
  Week 4 | 22.07 (14.342)
  Week 8: number analyzed (Participants) | 9
  Week 8 | 17.32 (8.042)
  Week 12 | 17.89 (9.646)
  Week 16 | 18.01 (10.610)
  Week 20 | 19.91 (15.436)
  Week 24: number analyzed (Participants) | 8
  Week 24 | 18.93 (6.538)

13. Secondary Outcome: Absolute Values of Ferritin at Baseline and Week 24
Description: Blood samples were collected from participants at defined time points for the assessment of iron indices. Absolute values of ferritin was reported.
Time Frame: Baseline, Week 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: microgram per liter (mcg/L)
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 8
microgram per liter (mcg/L)
  Baseline | 10.0 (5.90)
  Week 24 | 12.0 (7.86)

14. Secondary Outcome: Absolute Values of Magnesium, Total Cholesterol, and Triglycerides at Week 24
Description: Blood samples were collected from participants at defined time points for the assessment of magnesium, total cholesterol, and triglycerides. Absolute values of magnesium, total cholesterol, and triglycerides measured as mmol/L at baseline and Week 24 was reported.
Time Frame: Baseline, Week 24
Population: The safety analysis set included all enrolled participants who received the study drug. Here, "overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable for specified timepoints in categories.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 8
mmol/L
  Magnesium at Baseline: number analyzed (Participants) | 6
  Magnesium at Baseline | 0.793 (0.0381)
  Magnesium at Week 24 | 0.858 (0.0245)
  Total Cholesterol at Baseline: number analyzed (Participants) | 6
  Total Cholesterol at Baseline | 3.819 (0.8786)
  Total Cholesterol at Week 24 | 3.604 (0.3118)
  Triglycerides at Baseline: number analyzed (Participants) | 6
  Triglycerides at Baseline | 2.033 (0.7946)
  Triglycerides at Week 24 | 1.094 (0.3745)

15. Secondary Outcome: Change From Baseline in Alpha-1 Antitrypsin Levels in Stool at Week 12 and Week 24
Time Frame: Week 12, Week 24
Population: The FAS included all enrolled participants who received the study drug.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
milligrams per deciliter (mg/dL)
  Change from Baseline to Week 12: number analyzed (Participants) | 5
  Change from Baseline to Week 12 | -527.80 (318.818)
  Change from Baseline to Week 24: number analyzed (Participants) | 7
  Change from Baseline to Week 24 | -463.71 (204.250)

16. Secondary Outcome: Change From Baseline in Alpha-1 Antitrypsin Levels in Blood at Week 12 and Week 24
Time Frame: Week 12, Week 24
Population: Number of participants based on the total in the safety analysis set (SAF)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
mg/dL
  Change from Baseline to Week 12: number analyzed (Participants) | 8
  Change from Baseline to Week 12 | -57.8 (33.15)
  Change from Baseline to Week 24: number analyzed (Participants) | 9
  Change from Baseline to Week 24 | -43.4 (35.89)

17. Secondary Outcome: Percentage of Participants With Active Disease at Baseline Who Maintained Disease Control
Description: Measured by normalization of serum albumin, no worsening of facial or peripheral edema, increase in bowel movement, or increase in abdominal pain frequency, no increase in dose of permitted concomitant medication for the treatment of PLE at any time as described in the protocol
Time Frame: Weeks 12 to 48; Weeks 12 to 144; Weeks 24 to 48; Weeks 48 to 96; Weeks 96 to 144
Population: All enrolled participants who received the study drug. 1 participant was consented to Protocol Amendment 5, and completed the study at week 104. The remaining 9 participants were consented to Protocol Amendment 6 and completed the study at week 144.
Measure: Number; unit: percentage of participants
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
percentage of participants
  Weeks 12 to 48 | 100
  Weeks 12 to 144: number analyzed (Participants) | 9
  Weeks 12 to 144 | 100
  Weeks 24 to 48 | 100
  Weeks 48 to 96 | 100
  Weeks 96 to 144: number analyzed (Participants) | 9
  Weeks 96 to 144 | 100

18. Secondary Outcome: Change From Baseline in Physician Assessment of Facial Edema Based on a 5-point Likert Rating Scale
Description: The physician assessment of facial edema is based on a 5-point Likert scale ranging from no edema (1) to very severe edema (5).
Time Frame: Baseline and Week 144
Population: All enrolled participants who received the study drug and consented to Protocol Amendment 6 and who were evaluable at both time points for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 9
score on a scale | -1.7 (0.87)

19. Secondary Outcome: Change From Baseline in Physician Assessment of Peripheral Edema Based on a 5-point Likert Rating Scale
Description: The physician assessment of peripheral edema is based on a 5-point Likert scale ranging from no edema (1) to very severe edema (5).
Time Frame: Baseline and Week 144
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 9
score on a scale | -1.7 (0.71)

20. Secondary Outcome: Change From Baseline in Food and Drink Limitations as Assessed by the PedsQL™ GI Symptom Scales' Food and Drink Limits Sub-scale
Description: Frequency of limitations is assessed on a 5-point Likert response scale, ranging from never a problem (0) to almost always a problem (4). Items were reverse scored and linearly transformed to a 0 to 100 scale, where lower scores indicate more frequent problems with food and drink limitations.
Time Frame: Baseline and Week 144
Population: All enrolled participants who received the study drug and consented to Protocol Amendment 6 and who were evaluable at this time point for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 8
score on a scale | 47.40 (36.653)

21. Secondary Outcome: Change From Baseline in Health-Related Quality of Life (HRQoL) as Assessed by the PedsQL™ Generic Core Scales
Description: Physical functioning, emotional functioning, social functioning, and school/work/studies functioning is assessed using a 5-point Likert scale, ranging from never a problem (0) to almost always a problem (4). Items were reverse-scored and linearly transformed to a 0 to 100 scale, with higher scores indicating better HRQoL. The total scale score is computed as the sum of all the items over the number of items answered on individual scales. Subscale score is calculated as the sum of the items in the scale divided by the number of items answered in the scale.
Time Frame: Baseline and Week 144
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 8
score on a scale
  Week 144 Change from Baseline Total score of PedsQL Core Score | 26.55 (17.023)
  Week 144 Change from Baseline Subscale score: Physical functioning | 14.45 (39.900)
  Week 144 Change from Baseline Subscale score: Emotional functioning | 26.3 (28.88)
  Week 144 Change from Baseline Subscale score: Social functioning | 30.6 (20.43)
  Week 144 Change from Baseline Subscale score: School functioning: number analyzed (Participants) | 7
  Week 144 Change from Baseline Subscale score: School functioning | 41.43 (19.518)

22. Secondary Outcome: Number of Participants With Albumin Infusion by 24 Week Periods
Time Frame: Weeks 0 to 24; Weeks 24 to 48; Weeks 48 to 72; Weeks 72 to 96; Weeks 96 to 120; Weeks 120 to 144
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
Participants
  Weeks 0 to 24 | 1
  Weeks 24 to 48 | 0
  Weeks 48 to 72 | 0
  Weeks 72 to 96 | 0
  Weeks 96 to 120: number analyzed (Participants) | 9
  Weeks 96 to 120 | 0
  Weeks 120 to 144: number analyzed (Participants) | 9
  Weeks 120 to 144 | 0

23. Secondary Outcome: Change From Baseline in Albumin Values
Time Frame: Baseline and Week 144
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
grams per deciliter (g/dL) | 2.400 (0.6103)

24. Secondary Outcome: Percentage Change From Baseline in Albumin Values
Time Frame: Baseline and Week 144
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
percentage of change | 127.489 (81.0666)

25. Secondary Outcome: Time to First Normalization for Albumin Values
Time Frame: Baseline up to Week 144
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
days | 15.5 [8 to 28]

26. Secondary Outcome: Change From Baseline in Protein Values
Time Frame: Baseline and Week 144
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 8
grams per liter (g/L) | 37.13 (10.789)

27. Secondary Outcome: Time to First Normalization for Total Protein
Time Frame: Baseline up to Week 144
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
days | 22.0 [9 to 35]

28. Secondary Outcome: Change From Baseline in Immunoglobulin (Ig) Values
Time Frame: Baseline and Week 144
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 9
mg/dL | 1271.2 (261.91)

29. Secondary Outcome: Time to First Normalization for Ig Values
Time Frame: Baseline up to Week 144
Population: All enrolled participants with available Ig lab reference ranges.
Measure: Median (Full Range); unit: days
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 1
days | 341 [341 to 341]

30. Secondary Outcome: Change From Baseline in IgG Values
Time Frame: Baseline and Week 144
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 9
g/L | 10.626 (2.2486)

31. Secondary Outcome: Time to First Normalization for IgG Values
Time Frame: Baseline up to Week 144
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
days | 29.0 [8 to 29]

32. Secondary Outcome: Change From Baseline in IgM Values
Time Frame: Baseline and Week 144
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 9
mg/dL | 112.0 (51.21)

33. Secondary Outcome: Time to First Normalization for IgM Values
Time Frame: Baseline up to Week 44
Population: All enrolled participants who received the study drug who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: days
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 9
days | 1 [1 to 9]

34. Secondary Outcome: Change From Baseline in IgA Values
Time Frame: Baseline and Week 144
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 9
mg/dL | 96.7 (28.78)

35. Secondary Outcome: Time to First Normalization for IgA Values
Time Frame: Baseline up to Week 144
Measure: Median (Full Range); unit: days
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
days | 1 [1 to 9]

36. Secondary Outcome: Change From Baseline in Vitamin B12 Values
Time Frame: Baseline and Week 144
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: picomoles per liter (pmol/L)
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 6
picomoles per liter (pmol/L) | 138.8 (56.07)

37. Secondary Outcome: Time to First Normalization for Vitamin B12 Values
Time Frame: Baseline up to Week 144
Measure: Median (Full Range); unit: days
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
days | 8 [1 to 8]

38. Secondary Outcome: Change From Baseline in Vitamin B9 (Folate) Values
Time Frame: Baseline and Week 144
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: nanomole per liter (nmol/L)
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 6
nanomole per liter (nmol/L) | 2.92 (10.241)

39. Secondary Outcome: Time to First Normalization for Vitamin B9 (Folate) Values
Time Frame: Baseline up to Week 144
Measure: Median (Full Range); unit: days
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
days | 1 [1 to 8]

40. Secondary Outcome: Change From Baseline in Iron Values
Time Frame: Baseline and Week 144
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: micromole/liter (umol/L)
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 9
micromole/liter (umol/L) | 7.82 (4.091)

41. Secondary Outcome: Time to First Normalization for Iron Values
Time Frame: Baseline up to Week 144
Measure: Median (Full Range); unit: days
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
days | 97.5 [1 to 337]

42. Secondary Outcome: Change From Baseline in Unsaturated Iron Binding Capacity
Time Frame: Baseline and Week 144
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 8
umol/L | 16.20 (13.811)

43. Secondary Outcome: Time to First Normalization for Unsaturated Iron Binding Capacity
Time Frame: Baseline up to Week 144
Measure: Median (Full Range); unit: days
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
days | 1 [1 to 56]

44. Secondary Outcome: Change From Baseline in Ferritin Values
Time Frame: Baseline and Week 144
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: microgram per liter (ug/L)
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 6
microgram per liter (ug/L) | 32.0 (23.67)

45. Secondary Outcome: Time to First Normalization for Ferritin Values
Time Frame: Baseline up to Week 144
Measure: Median (Full Range); unit: days
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
days | 28 [1 to 505]

46. Secondary Outcome: Change From Baseline in Magnesium Values
Time Frame: Baseline and Week 144
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 6
millimoles per liter (mmol/L) | 0.083 (0.0606)

47. Secondary Outcome: Time to First Normalization for Magnesium Values
Time Frame: Baseline up to Week 144
Measure: Median (Full Range); unit: days
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
days | 1 [1 to 2]

48. Secondary Outcome: Change From Baseline in Fasting Cholesterol Values
Time Frame: Baseline and Week 144
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 6
mmol/L | -0.072 (0.7299)

49. Secondary Outcome: Time to First Normalization for Fasting Cholesterol Values
Time Frame: Baseline up to Week 144
Measure: Median (Full Range); unit: days
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
days | 1 [1 to 29]

50. Secondary Outcome: Change From Baseline in Fasting Triglycerides Values
Time Frame: Baseline and Week 144
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 6
mmol/L | -0.710 (0.9086)

51. Secondary Outcome: Time to First Normalization for Fasting Triglycerides Values
Time Frame: Baseline up to Week 144
Measure: Median (Full Range); unit: days
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
days | 4 [1 to 57]

52. Secondary Outcome: Number of Participants Who Used Concomitant Medication
Time Frame: Baseline up to Week 144
Measure: Count of Participants; unit: Participants
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
Participants | 10

53. Secondary Outcome: Number of Hospitalization Days by 24 Week Period
Time Frame: Weeks 0 to 24; Weeks 24 to 48; Weeks 48 to 72; Weeks 72 to 96; Weeks 96 to 120; Weeks 120 to 144
Population: All enrolled participants who received the study drug. 1 participant was consented to Protocol Amendment 5 and completed the study at week 104. The remaining 9 participants were consented to Protocol Amendment 6 and completed the study at week 144.
Measure: Median (Full Range); unit: days
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
days
  Weeks 0 to 24 | 0.0 [0 to 4]
  Weeks 24 to 48 | 0.0 [0 to 0]
  Weeks 48 to 72 | 0.0 [0 to 0]
  Weeks 72 to 96 | 0.0 [0 to 0]
  Weeks 96 to 120: number analyzed (Participants) | 9
  Weeks 96 to 120 | 0.0 [0 to 2]
  Weeks 120 to 144: number analyzed (Participants) | 9
  Weeks 120 to 144 | 0.0 [0 to 0]

54. Secondary Outcome: Change From Baseline in Body Weight Z-Score
Description: Weight-for-age z-score compares a participant's weight to children of the same age and sex from a healthy reference population. A z-score reflects an individual score as compared to a population mean and is expressed in units of standard deviation above (positive values) and below (negative values). Body weight z-score, regardless of magnitude, represents catch-up growth.
Time Frame: Baseline and Week 144
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 8
z-score | 0.924 (0.7529)

55. Secondary Outcome: Change From Baseline in Height Z-Score
Description: Height-for-age z-score compares a participant's height to children of the same age and sex from a healthy reference population. A z-score reflects an individual score as compared to a population mean and is expressed in units of standard deviation above (positive values) and below (negative values). Any increase in height z-score, regardless of magnitude, represents catch-up growth.
Time Frame: Baseline and Week 144
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 8
z-score | 1.079 (0.6469)

56. Secondary Outcome: Change From Baseline in Total Complement Activity Complement Hemolytic Assay (CH50)
Time Frame: Baseline and Week 144
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: international units/milliliter (IU/mL)
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 9
international units/milliliter (IU/mL) | -241.6 (39.79)

57. Secondary Outcome: Concentrations of Total Pozelimab in Serum
Time Frame: Baseline up to Week 164
Population: The Pharmacokinetic Analysis Set (PKAS) includes all treated participants who received any amount of study drug and had at least 1 non-missing total pozelimab measurement following the first dose of study drug. The PKAS is based on the actual treatment received (as treated) rather than as randomized.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
mg/L
  Week 1 | 182 (68.9)
  Week 2 | 185 (103)
  Week 4 | 227 (110)
  Week 6 | 268 (106)
  Week 8: number analyzed (Participants) | 9
  Week 8 | 306 (111)
  Week 12 | 341 (115)
  Week 16 | 402 (141)
  Week 20 | 418 (136)
  Week 24: number analyzed (Participants) | 8
  Week 24 | 421 (129)
  Week 36 | 467 (127)
  Week 48: number analyzed (Participants) | 9
  Week 48 | 517 (142)
  Week 72 | 492 (131)
  Week 96: number analyzed (Participants) | 9
  Week 96 | 461 (115)
  Week 144: number analyzed (Participants) | 9
  Week 144 | 430 (134)
  Week 145: number analyzed (Participants) | 1
  Week 145 | NA (NA) — Mean and Standard Deviation (SD) not calculable with n=1
  Week 146: number analyzed (Participants) | 1
  Week 146 | NA (NA) — Mean and Standard Deviation (SD) not calculable with n=1
  Week 164: number analyzed (Participants) | 8
  Week 164 | 410 (104)

58. Secondary Outcome: Number of Participants With Treatment-emergent Anti-drug Antibodies (ADA) to Pozelimab
Time Frame: Baseline up to Week 164
Population: The Anti-Drug Antibody Analysis Set (AAS) includes all treated participants who received any amount of study drug and had at least 1 non-missing ADA result following the first dose of study drug. The AAS is based on the actual treatment received (as treated) rather than as randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Pozelimab Injection
Number analyzed (Participants) | 10
Participants | 0

ADVERSE EVENTS:
Time Frame: From signing of informed consent up to 164 weeks (end of study)
Arm/Group | Pozelimab Injection
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 5/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pozelimab Injection (N=10)
Vomiting (Gastrointestinal disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pozelimab Injection (N=10)
Rhinitis (Infections and infestations) | 2 (2)
Acarodermatitis (Infections and infestations) | 2 (3)
Nasopharyngitis (Infections and infestations) | 3 (3)
Tonsillitis (Infections and infestations) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia areata (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (5)
Constipation (Gastrointestinal disorders) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4)
Pyrexia (General disorders) | 2 (3)
Hepatic enzyme increased (Investigations) | 1 (1)
Anaemia folate deficiency (Blood and lymphatic system disorders) | 1 (2)
Immunisation reaction (Immune system disorders) | 1 (3)
Headache (Nervous system disorders) | 2 (3)
Haematuria (Renal and urinary disorders) | 1 (3)
Proteinuria (Renal and urinary disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (6)
COVID-19 (Infections and infestations) | 2 (2)
Coronavirus infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (5)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1)
Folate deficiency (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)
Chronic spontaneous urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1)
Injection site erythema (General disorders) | 1 (3)
Oedema peripheral (General disorders) | 1 (1)
Xerosis (General disorders) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
"Blood 1,25-dihydroxycholecalciferol increased" (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Blood immunoglobulin M decreased (Investigations) | 1 (1)
Blood zinc decreased (Investigations) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Eyelid oedema (Eye disorders) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT04209634/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/34/NCT04209634/SAP_001.pdf